CLINICAL TRIAL: NCT01894087
Title: A Brief Prescription Opioid Overdose Intervention in an Emergency Department
Brief Title: Safety & Prevention Outcomes Study
Acronym: SPOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amy S.B. Bohnert, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R49CE002099 (NIH)
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Results first posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2017-05

CONDITIONS: Drug Overdose; Opioid-Related Disorders
MeSH Terms: conditions — Drug Overdose; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Therapist-led brief intervention (TBI) - Cohort 1 (Active Comparator): Participants will receive a therapist-led, computer-assisted intervention session with a master's level therapist. The interventions are designed to address extramedical prescription opioid use and overdose risk behaviors. This includes a review of the participants' strengths, values, and goals; feedback regarding their opioid use and overdose risk behaviors; developing a discrepancy between their opioid and other drug use and ability to meet goals and values; and the formulation of a "change plan" for each participant.
  Interventions: Behavioral: TBI - Cohort 1
- Enhanced usual care - Cohort 1 (No Intervention)
- Therapist-led brief intervention (TBI) - Cohort 2 (Active Comparator): Participants will receive a therapist-led, computer-assisted intervention session with a master's level therapist. The interventions are designed to address extramedical prescription opioid use and overdose risk behaviors. This includes a review of the participants' strengths, values, and goals; feedback regarding their opioid use and overdose risk behaviors; developing a discrepancy between their opioid and other drug use and ability to meet goals and values; and the formulation of a "change plan" for each participant.
  Interventions: Behavioral: TBI - Cohort 2
- Enhanced usual care - Cohort 2 (No Intervention)

INTERVENTIONS:
Behavioral: TBI - Cohort 1
  Arms: Therapist-led brief intervention (TBI) - Cohort 1
Behavioral: TBI - Cohort 2
  Arms: Therapist-led brief intervention (TBI) - Cohort 2

SUMMARY:
Unintentional poisoning is a developing public health problem in the U.S. Unintentional poisoning (or "overdose") deaths increased 157% among adults between 1999 and 2008. There were ~700,000 emergency department (ED) visits due to overdoses in 2007. Medication-related overdoses, particularly prescription opioid overdoses, have accounted for much of this increase. There have been parallel increases in sales of opioids (with a 6 fold increase between 1997 and 2007), as well as both medical and non-medical use of prescription opioids. Prescription opioids are now among the most common of drugs used non-medically in the U.S.

The specific aims of this project are to: 1) Develop an ED-based tailored brief prescription opioid overdose prevention intervention. We will examine therapeutic alliance, perceived satisfaction, and perceived utility of the intervention; 2) Examine intervention effects on precursors of overdose risk behavioral change immediately post-intervention. We will compare intervention and control participants on knowledge, self-efficacy, readiness to change, and behavioral intentions regarding overdose risk behavior; and 3) Examine intervention effects on overdose risk behaviors six months post-intervention. We will compare intervention and control participants on: 1) use of high dose/quantity of opioids; 2) using opioids in combinations with certain psychoactive substances (i.e., alcohol, heroin, cocaine, and sedatives); and, 3) route of administration.

ELIGIBILITY:
Inclusion Criteria:

* patients 18-60 presenting to the ED for medical care
* ability to provide informed consent
* Additional criteria for intervention: past extramedical opioid use

Exclusion Criteria:

* patients who do not understand English
* prisoners
* patients classified by medical staff as a "Level 1" trauma (e.g., in need of immediate lifesaving procedures)
* patients deemed unable to provide informed consent
* patients treated in the ED for suicide attempt or sexual assault

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Bohnert, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System Emergency Department, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Bohnert AS, Bonar EE, Cunningham R, Greenwald MK, Thomas L, Chermack S, Blow FC, Walton M. A pilot randomized clinical trial of an intervention to reduce overdose risk behaviors among emergency department patients at risk for prescription opioid overdose. Drug Alcohol Depend. 2016 Jun 1;163:40-7. doi: 10.1016/j.drugalcdep.2016.03.018. Epub 2016 Mar 26. PMID 27062245

RESULTS

PARTICIPANT FLOW:
Groups:
- Therapist-led Brief Intervention With Enhanced Usual Care: Participants will receive a therapist-led, computer-assisted intervention session with a master's level therapist. The interventions are designed to address extramedical prescription opioid use and overdose risk behaviors. This includes a review of the participants' strengths, values, and goals; feedback regarding their opioid use and overdose risk behaviors; developing a discrepancy between their opioid and other drug use and ability to meet goals and values; and the formulation of a "change plan" for each participant. Participants in this condition also received the brochures given for the Enhanced Usual Care protocol.
- Enhanced Usual Care Only: For Enhanced Usual Care (EUC), therapists provided two brochures: (1) an overdose prevention and response brochure, and (2) a resource brochure. The overdose prevention and response brochure included a definition of overdose, signs and symptoms, risk factors, and bystander response to overdose. The resource brochure contained information on drug,mental health and alcohol treatment, mutual help groups, local resources for obtaining naloxone, free health clinics in the area, and a suicide prevention hotline.
Period: Overall Study
Arm/Group | Therapist-led Brief Intervention With Enhanced Usual Care | Enhanced Usual Care Only
Started | 102 | 102
Completed | 96 | 102
Not Completed | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Therapist-led Brief Intervention With Enhanced Usual Care | Enhanced Usual Care Only | Total
Number analyzed (Participants) | 102 | 102 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (11.4) | 36.1 (10.9) | 36.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 69 | 130
  Male | 41 | 33 | 74
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 69 | 79 | 148
  Black | 22 | 16 | 38
  Other/Missing/More than 1 | 11 | 7 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 102 | 102 | 204

OUTCOME MEASURES:

1. Primary Outcome: Overdose Risk Behavior
Description: This scale is a total sum of 9 items assessing participant's self-report of engaging in behavior that increases risk for overdose. Higher scores indicate greater risk for overdose. The range for this measure is 0 to 28 in one assessment. Results reported here as group means are for the change in sum score between baseline and follow-up, which had a possible range of -28 to 28, with lower values indicating greater decreases in overdose risk behavior.
Time Frame: 6 months post-baseline
Population: Participants who were retained at follow-up and had complete data for all items for this measure at baseline and follow-up
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Therapist-led Brief Intervention With Enhanced Usual Care | Enhanced Usual Care Only
Number analyzed (Participants) | 92 | 80
Scores on a scale | -1.54 [-2.57 to -0.52] | -0.51 [-1.75 to 0.72]
Statistical Analysis 1: Comparison: Therapist-led Brief Intervention With Enhanced Usual Care vs Enhanced Usual Care Only; Multivariable Poisson regression of outcome of overdose risk behavior sum score at 6 months, adjusting for baseline level of the outcome; Test type: Superiority; Incidence Rate Ratio = 0.72, 95% CI 2-sided [0.59 to 0.87] — Numerator is Therapist-led Brief Intervention, Denominator is Enhanced Usual Care only

2. Primary Outcome: Overdose Knowledge
Description: Overdose symptom knowledge was assessed using an inventory of 5 true symptoms and 2 false symptoms of overdose, and the total score created as the sum of correct answers, with a range of 0 to 7. Due to the skewed distribution, this total score was standardized by subtracting the observed responses from the overall sample mean, and then dividing by the standard deviation. This resulted in a range of -5.4 to 2.6 in this sample at the 6 month follow-up, with higher numbers indicating greater overdose symptom knowledge. Also reported here are change scores generated by subtracting the standardized sum score at 6 months from the baseline standardized sum score, which had a range of -3.0 to 6.4 in this sample. Thus, higher numbers in this "change" variable indicated greater improvements in overdose symptom knowledge. Negative numbers would represent a decrease in symptom knowledge.
Time Frame: 6 months post-baseline
Population: Participants retained and follow-up and with complete data on the outcome measure items at baseline and follow-up.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Therapist-led Brief Intervention With Enhanced Usual Care | Enhanced Usual Care Only
Number analyzed (Participants) | 91 | 81
Scores on a scale | 0.12 [-0.12 to 0.36] | -0.11 [-0.41 to 0.18]
Statistical Analysis 1: Comparison: Therapist-led Brief Intervention With Enhanced Usual Care vs Enhanced Usual Care Only; Multivariable linear regression of the outcome of standardized sum score of overdose symptom knowledge at 6 months follow-up, adjusted for baseline level of overdose symptom knowledge; Test type: Superiority; Slope = 0.10, 95% CI 2-sided [-0.20 to 0.40] — Numerator is the Therapist-Led Brief Intervention and Denominator is Enhanced Usual Care only

3. Primary Outcome: Behavioral Intentions
Description: Behavioral intentions were assessed with three items that measured participant's intention to use overdose risk reduction strategies. The three strategies were (1) using opioids as prescribed, (2) reducing or avoiding use of alcohol, drugs, or non-prescribed medications, and (3) avoiding combining substances. Each item was assessed on a scale of 1 to 10, with higher numbers indicating greater intention to avoid overdose risk.
Time Frame: 6 months post-baseline
Population: Participants retained at follow-up and with complete item data on the outcome at baseline and follow-up
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Therapist-led Brief Intervention With Enhanced Usual Care | Enhanced Usual Care Only
Number analyzed (Participants) | 88 | 80
Scores on a scale
  Use opioids as prescribed | 8.0 [7.4 to 8.6] | 8.4 [7.8 to 8.9]
  Reducing or avoiding all use | 8.1 [7.5 to 8.6] | 7.0 [6.3 to 7.8]
  Avoid combining substances | 8.7 [8.2 to 9.3] | 8.6 [8.0 to 9.2]
Statistical Analysis 1: Comparison: Therapist-led Brief Intervention With Enhanced Usual Care vs Enhanced Usual Care Only; Multivariable Poisson regression of the outcome of intention to use opioids as prescribed, adjusting for baseline level of the outcome; Test type: Superiority; Incidence Rate Ratio = 1.11, 95% CI 2-sided [0.93 to 1.33] — This item was reverse coded; higher scores indicate lower intention to avoid overdose risk (for the strategy of using opioids as prescribed). Numerator was the Therapist-Led Brief Intervention and the denominator was Enhanced Usual Care only
Statistical Analysis 2: Comparison: Therapist-led Brief Intervention With Enhanced Usual Care vs Enhanced Usual Care Only; Multivariable Poisson regression of the outcome of intention to avoid or reduce opioid use, adjusting for baseline level of the outcome; Test type: Superiority; Incidence Rate Ratio = 0.76, 95% CI 2-sided [0.65 to 0.90] — This item was reverse coded; higher scores indicate lower intention to avoid overdose risk (for the strategy of reducing or avoiding opioid use). Numerator was the Therapist-Led Brief Intervention and the denominator was Enhanced Usual Care only
Statistical Analysis 3: Comparison: Therapist-led Brief Intervention With Enhanced Usual Care vs Enhanced Usual Care Only; Multivariable Poisson regression of the outcome of intention to avoid combining opioids with other substances, adjusting for baseline level of the outcome; Test type: Superiority; Incidence Rate Ratio = 0.97, 95% CI 2-sided [0.80 to 1.19] — This item was reverse coded; higher scores indicate lower intention to avoid overdose risk (for the strategy of not combining opioids with other drugs). Numerator was Therapist-Led Brief Intervention and denominator was Enhanced Usual Care only

4. Secondary Outcome: Substance Use - Current Opioid Misuse Measure
Description: This measure contained 8 items from the Current Opioid Misuse Measure. Items were assessed on a scale of "never (0)," "rarely (1)," "sometimes (3)," "often (4)," and "very often (5)." A sum score took a range of 0 to 40, with higher numbers indicating more non-medical opioid use. For group means reported here, change scores were calculated by subtracting the baseline level of this measure from the level at 6 months follow-up. This change score has a possible range of -40 to 40, with lower values indicating greater decreases in non-medical opioid use.
Time Frame: 6 months post-baseline
Population: Participants retained at follow-up and with complete item data on this measure at both baseline and follow-up
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Therapist-led Brief Intervention With Enhanced Usual Care | Enhanced Usual Care Only
Number analyzed (Participants) | 87 | 76
Scores on a scale | -4.44 [-6.41 to -2.47] | -3.54 [-5.84 to -1.24]
Statistical Analysis 1: Comparison: Therapist-led Brief Intervention With Enhanced Usual Care vs Enhanced Usual Care Only; Multivariable Poisson regression for the outcome of total COMM score at follow-up, adjusting for baseline level of the outcome; Test type: Superiority; Incidence Rate Ratio = 0.81, 95% CI 2-sided [0.70 to 0.92] — Numerator is Therapist-Led Brief Intervention, Denominator is Enhanced Usual Care only

ADVERSE EVENTS:
Arm/Group | Therapist-led Brief Intervention With Enhanced Usual Care | Enhanced Usual Care Only
All-Cause Mortality (participants affected / at risk) | 1/102 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/102
Other Adverse Events (participants affected / at risk) | 0/102 | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No